CLINICAL TRIAL: NCT00619983
Title: Three Way Interaction Between Gabapentin, Duloxetine, and Donepezil in Patients With Diabetic Neuropathy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to low enrollment
Sponsor: Wake Forest University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00003943; 5R01NS057594 (NIH)
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Diabetic Neuropathic Pain; Chronic Low Back Pain
Keywords: Asymmetric Diabetic Proximal Motor Neuropathy; Diabetic Autonomic Neuropathy; Diabetic Neuralgia; Diabetic Neuropathy, Painful; Neuralgia, Diabetic; Low back pain, chronic
MeSH Terms: conditions — Diabetic Neuropathies; Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Donepezil; Duloxetine Hydrochloride; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Donepezil (Active Comparator): Donepezil 5 mg once per day for 12 weeks. Gabapentin will be titrated in all groups beginning at week 8.
  Interventions: Drug: donepezil; Drug: gabapentin
- Duloxetine (Active Comparator): Group 2: Will receive duloxetine 30 mg twice a day for 12 weeks. Gabapentin will be titrated in all groups beginning at week 8.
  Interventions: Drug: duloxetine; Drug: gabapentin
- Donepezil + Duloxetine (Active Comparator): Group 3: Will receive a combination of donepezil 2.5 mg and duloxetine 30mg for 12 weeks. Gabapentin will be titrated in all groups beginning at week 8.
  Interventions: Drug: donepezil 2.5 mg and duloxetine 30mg; Drug: gabapentin
- Placebo (Placebo Comparator): Group 4:Will receive placebo pills. Gabapentin will be titrated in all groups beginning at week 8.
  Interventions: Drug: placebo; Drug: gabapentin

INTERVENTIONS:
Drug: donepezil — Group 1: Will receive donepezil 5mg once a day
  Other Names: Aricept®
  Arms: Donepezil
Drug: duloxetine — Group 2: Will receive duloxetine 30 mg twice a day
  Other Names: Cymbalta®
  Arms: Duloxetine
Drug: donepezil 2.5 mg and duloxetine 30mg — Group 3: Will receive a combination of donepezil 2.5 mg and duloxetine 30mg
  Other Names: Cymbalta®; Aricept®
  Arms: Donepezil + Duloxetine
Drug: placebo — Group 4: Will receive placebo pills
  Arms: Placebo
Drug: gabapentin — Week 8: all subjects will have open label gabapentin added to their randomized study medication
  Other Names: neurontin

SUMMARY:
The purpose of the study is to determine whether the combination of the the three drugs gabapentin, duloxetine, and donepezil are effective in treating pain in people with diabetic neuropathy or patients with failed low back syndrome (chronic back pain).

DETAILED DESCRIPTION:
Neuropathic pain is a complex and likely heterogeneous disorder, and we recognize that clinically useful agents such as opioids, gabapentin, and antidepressants may be effective precisely because they have multiple mechanisms of action at multiple sites. This study, however, will not only provide important mechanistic information regarding one cascade which can be manipulated for analgesia, but will also provide much needed systematic and practical guidance for multi-drug therapy in patients with neuropathic pain.

This study in patients with diabetic neuropathic pain and patients with failed low back syndrome, culminate in a quantitative description of interactions between activators of descending noradrenergic activity, norepinephrine transporter inhibitors, and cholinesterase inhibitors to exploit the plasticity of analgesia in chronic pain states. We will focus on practical applications, using clinically approved drugs, including gabapentin (Neurontin®) to activate noradrenergic activity, duloxetine (Cymbalta®) to inhibit the norepinephrine transporter, and donepezil (Aricept®), approved for the treatment of Alzheimer's dementia, but not previously tested to treat neuropathic pain, to inhibit cholinesterase.

After the baseline measurements and physical examination patients will be trained to use a Personal Digital Assistant (PDA) to answer questions about their diabetic neuropathic pain or their chronic back pain. Upon successful completion of these tasks the patients will be randomized to receive one of the drug choices or placebo (inactive pill).

The study will last for a total of 16 weeks and includes 5 visits to the research center with each visit lasting approximately 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetic neuropathy
* Age 18-80
* Willing to temporarily discontinue gabapentin or monoamine reuptake inhibitors upon entry into the study

Exclusion Criteria:

* Pregnancy
* Allergy to study medications
* Uncontrolled narrow-angle glaucoma
* Currently being treatment with thioridazine (Mellaril)
* Unstable medical conditions including cardiac, pulmonary, renal or hepatic diseases
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 days of randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
Raw IPD will not be shared

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil: Donepezil 5 mg /day from 2-14 weeks with gabapentin titrated beginning at week 8 and maintained until week 15.
- Duloxetine: Duloxetine 30 mg twice per day from 2-14 weeks with gabapentin titrated beginning at week 8 and maintained until week 15.
- Donepezil + Duloxetine: Donepezil 2.5 mg /day and duloxetine 30 mg / day from 2-14 weeks with gabapentin titrated beginning at week 8 and maintained until week 15.
- Placebo: Placebo from 2-14 weeks with gabapentin titrated beginning at week 8 and maintained until week 15.
Period: Test Drug Alone
Arm/Group | Donepezil | Duloxetine | Donepezil + Duloxetine | Placebo
Started | 5 | 5 | 6 | 6
Completed | 3 | 4 | 4 | 3
Not Completed | 2 | 1 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Failure of daily diary device | 1 | 1 | 2 | 2
Period: Test Drug Plus Gabapentin
Arm/Group | Donepezil | Duloxetine | Donepezil + Duloxetine | Placebo
Started | 3 | 4 | 4 | 3
Completed | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Gabapentin Alone
Arm/Group | Donepezil | Duloxetine | Donepezil + Duloxetine | Placebo
Started | 3 | 4 | 4 | 3
Completed | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Duloxetine | Donepezil + Duloxetine | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 6 | 6 | 22
Age, Continuous [Median (Full Range); unit: years] | 62 [52 to 65] | 56 [54 to 60] | 59 [58 to 59] | 70 [65 to 72] | 60 [50 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 1 | 3 | 8
  Male | 1 | 5 | 5 | 3 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 1 | 7
  White | 3 | 3 | 4 | 5 | 15
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 6 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale for Pain
Description: The primary outcome measure is the visual analog scale (VAS) for pain, a 10 cm line upon which the subject marks their intensity of pain. The line is anchored on the left as "No pain at all" and on the right as "The worst pain imaginable". The score is the number of millimeters from the left origin of the line. The primary outcome measure for each period was the average value of all assessments for that period (2 weeks of measures for baseline, 6 weeks of measures for test drug alone, 6 weeks of measures for test drug plus gabapentin, and 2 weeks of measures for gabapentin alone).
Time Frame: Study completion (16 weeks)
Population: As noted in patient flow, data are available for only 14 of 22 subjects due to failure of the electronic daily diaries used to assess pain during the study and to study discontinuation in some cases
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Donepezil | Duloxetine | Donepezil + Duloxetine | Placebo
Number analyzed (Participants) | 3 | 4 | 4 | 3
units on a scale
  Baseilne ( weeks) | 3.3 [2.0 to 6.7] | 6.4 [2.3 to 9.8] | 5.8 [3.6 to 7.3] | 4.9 [4.5 to 8.4]
  Test drug alone (6 weeks) | 4.1 [1.5 to 4.6] | 2.9 [1.6 to 9.7] | 5.2 [4.3 to 6.9] | 3.9 [2.4 to 4.8]
  Drug plus gabapentin (6 weeks) | 2.9 [0.4 to 3.2] | 2.7 [1.1 to 9.7] | 3.9 [3.5 to 5.3] | 4.1 [1.1 to 6.3]
  Gabapentin alone (2 weeks) | 2.2 [0 to 2.6] | 3.0 [2.4 to 10] | 4.3 [3.3 to 5.2] | 4.1 [1.9 to 6.4]
Statistical Analysis 1: Comparison: Donepezil vs Duloxetine vs Donepezil + Duloxetine vs Placebo; Due to failure of daily electronic diaries and exhaustion of funds, we were only able to recruit < 30% of the number of subjects required in our power analysis; Test type: Superiority; p = 0.69, ANOVA; Repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: During the 16 week study
Arm/Group | Donepezil | Duloxetine | Donepezil + Duloxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 1/5 | 0/5 | 0/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=5) | Duloxetine (N=5) | Donepezil + Duloxetine (N=6) | Placebo (N=6)
Angina (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Subject experienced chest pain and was hospitalized. Serial ECGs and troponins were negative for myocardial injury
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=5) | Duloxetine (N=5) | Donepezil + Duloxetine (N=6) | Placebo (N=6)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — subject experienced nausea
osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — subject experienced osteomyelitis of of second phalange

LIMITATIONS AND CAVEATS:
We recruited only a small proportion of the planned enrollment in the period of grant funding, leading to early termination of the study. Also, the failure of the electronic diaries and loss of primary outcome data prevented the planned analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-10-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT00619983/Prot_SAP_000.pdf
  • Informed Consent Form (2010-04-16): https://cdn.clinicaltrials.gov/large-docs/83/NCT00619983/ICF_001.pdf